CLINICAL TRIAL: NCT02563964
Title: Characterizing Vulnerable Plaques in Non-ST-Elevation Myocardial Infarction Using 18F-NaF Positron Emission Tomography - Cardiac Magnetic Resonance Imaging: A Feasibility Study
Brief Title: Vulnerable Plaque Imaging in NSTEMI
Acronym: CULPRIT
Status: Terminated | Type: Observational
Why Stopped: Logistical reasons and slow recruitment
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL51875.068.14 / METC 152007
Record Dates: First submitted 2015-09-25; First posted 2015-09-30 (Estimated); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Myocardial Infarction; Myocardial Ischemia
Keywords: Myocardial infarction; vulnerable plaque; Positron emission tomography (PET); Cardiac magnetic resonance imaging (CMR); Biomarkers
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Biomarkers
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Myocardial infarction (MI) frequently recurs after non-ST elevation MI (NSTEMI) that may be related to insufficient vulnerable plaque identification using invasive coronary angiography. Furthermore, the natural behaviour of vulnerable plaques in NSTEMI over time and their relation with biomarkers need further exploration. More accurate identification and assessing long-term behaviour of vulnerable plaques may improve therapeutic strategies and clinical outcome. The investigators hypothesize that fully integrated 18Fluoride Sodium-Fluoride (18F-NaF) Positron Emission Tomography/Cardiac Magnetic Resonance imaging (PET/CMR) increases the ability to detect vulnerable plaques as compared to coronary angiography.

This prospective study in 33 consecutive patients with NSTEMI aims to:

1. Compare coronary vulnerable plaque detection between 18F-NaF PET/CMR and invasive coronary angiography,
2. Investigate the correlation of coronary vulnerable plaques using 18F-NaF PET with myocardial infarction using CMR, both at baseline and during follow-up,
3. Examine systemic arterial 18F-NaF-uptake using PET/CMR and their relation with systemic events (cerebrovascular accidents, transient ischemic attacks, or peripheral arterial disease), and
4. Examine the relation between vulnerable plaques and plasma biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Prolonged symptoms suspected of cardiac origin (angina pectoris or angina equivalent), and presentation on the cardiac emergency department <24 hours after symptom onset
* Elevated levels of high-sensitivity troponin T (>14ng/L; initial blood sample at presentation or a second sample 3 hours after presentation)
* Only patients scheduled for invasive coronary angiography
* Age 18 years - 85 years
* Mentally competent
* Informed written consent

Exclusion Criteria:

* Conservatively managed patients who are not scheduled for invasive coronary angiography
* Refractory angina or on-going severe ischemia requiring immediate invasive coronary angiography
* Patients requiring invasive coronary angiography < 24 hours after admission
* Hemodynamic instability and cardiogenic shock (mean arterial pressure < 60 mmHg)
* Severe heart failure (Killip Class ≥ III)
* ST elevation myocardial infarction (ST-elevation in 2 contiguous leads: ≥0.2mV in men or ≥0.15 mV in women in leads V2-V3 and/or ≥0.1 mV in other leads or new left bundle branch block)
* Chest pain highly suggestive of non-cardiac origin (as judged by the cardiac emergency department physician/cardiologist):
* (Suspicion of) acute aortic dissection, acute pulmonary embolism, acute peri-myocarditis
* Life threatening arrhythmias on the cardiac emergency department or prior to presentation (sustained ventricular tachycardia, repetitive non-sustained ventricular tachycardia, ventricular fibrillation, sino-artial or atrio-ventricular block)
* Atrial fibrillation with ventricular rate ≥100 beats per minute (bpm)
* Tachycardia (≥100/bpm)
* Angina pectoris secondary to anaemia (<5.6 mmol/L), untreated hyperthyroidism, or severe hypertension (>200/110 mmHg)
* More than mild aortic and mitral valve calcification or stenosis by latest echocardiography
* Pregnancy
* Breast feeding women
* Life expectancy <2 years (malignancy, etc.)
* Refusal of data storage until 15 years after end of study
* Participation in another investigational study that has not reached its primary endpoint
* Contraindications to cardiac magnetic resonance imaging

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty-three patients, 18-85 years old and admitted with non-ST elevation myocardial infarction (NSTEMI). After informed consent, patients wil receive standard, guideline-based clinical care that includes invasive coronary angiography. Plasma biomaker will be sampled serially, and a comprehensive Sodium 18F-Fluoride Positron Emission Tomography/Cardiac Magnetic Resonance imaging (18F-NaF PET/CMR) will be performed at baseline (<72 hours) and at 6 months, or earlier when patients suffer recurrent myocardial infarction < 6months. Patients will be followed for one year during regular outpatient clinic visits.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
The frequency of coronary vulnerable plaques in non-ST-elevation myocardial infarction (NSTEMI) using 18Fluoride Sodium-Fluoride (18F-NaF) Positron Emission Tomography/Cardiac Magnetic Resonance (PET/CMR). | 0 to 6 months
The frequency of coronary vulnerable plaques in NSTEMI using routine invasive coronary angiography. | 0 to 6 months

SECONDARY OUTCOMES:
The location of vulnerable plaques within the coronary arteries using 18F-NaF PET at baseline and follow-up. | 0 to 6 months
Based on the AHA 17-segment model, the segmental location of MI using CMR at baseline and follow-up. | 0 to 6 months
The frequency of systemic vulnerable plaques as assessed with 18F-NaF PET/CMR at baseline and follow-up. | 0 to 6 months
Serial serum concentrations of biomarkers of plaque vulnerability and myocardial injury at baseline and follow-up. | 0 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Wildberger, MD, PhD, Principal Investigator — Maastricht University Medical Center; Harry J. Crijns, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Libby P, Theroux P. Pathophysiology of coronary artery disease. Circulation. 2005 Jun 28;111(25):3481-8. doi: 10.1161/CIRCULATIONAHA.105.537878. PMID 15983262
- [Background] Virmani R, Kolodgie FD, Burke AP, Farb A, Schwartz SM. Lessons from sudden coronary death: a comprehensive morphological classification scheme for atherosclerotic lesions. Arterioscler Thromb Vasc Biol. 2000 May;20(5):1262-75. doi: 10.1161/01.atv.20.5.1262. No abstract available. PMID 10807742
- [Background] Cutlip DE, Chhabra AG, Baim DS, Chauhan MS, Marulkar S, Massaro J, Bakhai A, Cohen DJ, Kuntz RE, Ho KK. Beyond restenosis: five-year clinical outcomes from second-generation coronary stent trials. Circulation. 2004 Sep 7;110(10):1226-30. doi: 10.1161/01.CIR.0000140721.27004.4B. Epub 2004 Aug 30. PMID 15337693
- [Background] Glaser R, Selzer F, Faxon DP, Laskey WK, Cohen HA, Slater J, Detre KM, Wilensky RL. Clinical progression of incidental, asymptomatic lesions discovered during culprit vessel coronary intervention. Circulation. 2005 Jan 18;111(2):143-9. doi: 10.1161/01.CIR.0000150335.01285.12. Epub 2004 Dec 27. PMID 15623544
- [Background] Kim HW, Klem I, Shah DJ, Wu E, Meyers SN, Parker MA, Crowley AL, Bonow RO, Judd RM, Kim RJ. Unrecognized non-Q-wave myocardial infarction: prevalence and prognostic significance in patients with suspected coronary disease. PLoS Med. 2009 Apr 21;6(4):e1000057. doi: 10.1371/journal.pmed.1000057. Epub 2009 Apr 21. PMID 19381280
- [Background] Kato K, Yonetsu T, Kim SJ, Xing L, Lee H, McNulty I, Yeh RW, Sakhuja R, Zhang S, Uemura S, Yu B, Mizuno K, Jang IK. Nonculprit plaques in patients with acute coronary syndromes have more vulnerable features compared with those with non-acute coronary syndromes: a 3-vessel optical coherence tomography study. Circ Cardiovasc Imaging. 2012 Jul;5(4):433-40. doi: 10.1161/CIRCIMAGING.112.973701. Epub 2012 Jun 7. PMID 22679059
- [Background] Stone GW, Maehara A, Lansky AJ, de Bruyne B, Cristea E, Mintz GS, Mehran R, McPherson J, Farhat N, Marso SP, Parise H, Templin B, White R, Zhang Z, Serruys PW; PROSPECT Investigators. A prospective natural-history study of coronary atherosclerosis. N Engl J Med. 2011 Jan 20;364(3):226-35. doi: 10.1056/NEJMoa1002358. PMID 21247313
- [Background] Joshi NV, Vesey AT, Williams MC, Shah AS, Calvert PA, Craighead FH, Yeoh SE, Wallace W, Salter D, Fletcher AM, van Beek EJ, Flapan AD, Uren NG, Behan MW, Cruden NL, Mills NL, Fox KA, Rudd JH, Dweck MR, Newby DE. 18F-fluoride positron emission tomography for identification of ruptured and high-risk coronary atherosclerotic plaques: a prospective clinical trial. Lancet. 2014 Feb 22;383(9918):705-13. doi: 10.1016/S0140-6736(13)61754-7. Epub 2013 Nov 11. PMID 24224999
- [Background] Dweck MR, Chow MW, Joshi NV, Williams MC, Jones C, Fletcher AM, Richardson H, White A, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Coronary arterial 18F-sodium fluoride uptake: a novel marker of plaque biology. J Am Coll Cardiol. 2012 Apr 24;59(17):1539-48. doi: 10.1016/j.jacc.2011.12.037. PMID 22516444
- [Background] Kim RJ, Chen EL, Lima JA, Judd RM. Myocardial Gd-DTPA kinetics determine MRI contrast enhancement and reflect the extent and severity of myocardial injury after acute reperfused infarction. Circulation. 1996 Dec 15;94(12):3318-26. doi: 10.1161/01.cir.94.12.3318. PMID 8989146
- [Background] Kwee RM, van Oostenbrugge RJ, Mess WH, Prins MH, van der Geest RJ, ter Berg JW, Franke CL, Korten AG, Meems BJ, van Engelshoven JM, Wildberger JE, Kooi ME. MRI of carotid atherosclerosis to identify TIA and stroke patients who are at risk of a recurrence. J Magn Reson Imaging. 2013 May;37(5):1189-94. doi: 10.1002/jmri.23918. Epub 2012 Nov 16. PMID 23166040
- [Background] Ambrose JA, Winters SL, Stern A, Eng A, Teichholz LE, Gorlin R, Fuster V. Angiographic morphology and the pathogenesis of unstable angina pectoris. J Am Coll Cardiol. 1985 Mar;5(3):609-16. doi: 10.1016/s0735-1097(85)80384-3. PMID 3973257